CLINICAL TRIAL: NCT01179464
Title: Effect of Aminobiphosphonates and Statins on Circulating Vgamma9Vdelta2-T Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: H.M.W. Verheul, MD, PhD, Professor of Medical Oncology, VU University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/70
Record Dates: First submitted 2010-08-04; First posted 2010-08-11 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-05

CONDITIONS: Bone Metastases of a Malignant Tumor
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aminobiphosphonates (Active Comparator): Aminobiphosphonates
  Interventions: Drug: Aminobiphosphonate
- Aminobiphosphonates and Statin (Experimental): Aminobiphosphonates and Statin
  Interventions: Drug: Aminobiphosphonate; Drug: Simvastatin

INTERVENTIONS:
Drug: Aminobiphosphonate — Patients will receive standard intravenous biphosphonate treatment
Drug: Simvastatin — 40 mg once daily
  Arms: Aminobiphosphonates and Statin

SUMMARY:
The purpose of this study is to investigate the effects of aminobiphosphonate treatment on the phenotype and function of circulating Vgamma9Vdelta2-T cells and to determine whether these effects are inhibited by simultaneous treatment with statins.

DETAILED DESCRIPTION:
A total of 40 patients will be entered in this study. Half of the patients will receive standard intravenous treatment with aminobsiphosphonates, the other half will be additionally be treated with a statin. Patients already receiving statin treatment will continue this treatment, other patients will be asked whether they are willing to be treated with a statin for a maximum of 5 weeks. Consenting patients will be randomized to receive i.v. aminobisphosponates plus or minus simvastatin 40 mg once daily. Simvastatin will be started one week prior to the first administration of aminobisphosphonates and continued for a maximum of 5 weeks. In each patient 10 ml peripheral blood will be drawn (t=0, t=24 hr, t=1 week, t=3-4 weeks (prior to the 2nd aminobisphosphonate administration). In addition, patients will be requested to measure their temperature thrice daily during the 2 days following the first aminobisphosponate administration. This, because a relation between the occurrence of a febrile response upon aminobisphosponate administration and an activation and expansion of Vy9Vd2-T cells has been suggested. Peripheral blood mononuclear cells will be isolated from the drawn peripheral blood. Using intra- and extracellular flowcytometry Vy9Vd2-T cells will be characterized phenotypically (APC markers: CD1d, CD40, CD80, CD83, CD86, HLA-DR; activation/memory markers: CD25, CD27, CD45RA, CD45RO, CCR7) and functionally (IFN-γ, TNF-α, granzyme B). In addition, the frequency of CD3+, CD4+, CD8+ T cells, NK cells, B cells, iNKT cells, CD4+CD25+ regulatory T cells, and circulating dendritic cells will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for intravenous treatment with an aminobiphosphonate because of a malignant tumor
* WHO 0,1,2 performance score

Exclusion Criteria:

* WHO 3, 4 performance score
* prior or current use of aminobisphosphonates -immunosuppressive medication (NSAID allowed)
* chemotherapy and/or radiotherapy in 4 weeks prior to start of aminobisphosphonate administration
* renal insufficiency (creatinine clearance < 30 ml/min)
* liver enzyme abnormalities:

  * bilirubin > 1.5 times ULN (upper limit of normal)
  * ASAT or ALAT > 2.5 times ULN (in absence of liver metastases)
  * ASAT or ALAT > 5 times ULN (in presence of liver metastases)
* concomitant use of strong inhibitors of CYP3A4, such as itraconazole, ketoconazole, erytromycin, clarithromycin, hiv-protease inhibitors or grapefruit juice is contra-indicated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Phenotypic (APC markers: CD1d, CD40, CD80, CD83, CD86, HLA-DR; activation/memory markers: CD25, CD27, CD45RA, CD45RO, CCR7)changes in the circulating pool of Vy9Vd2-T cells. | 5 weeks
  Peripheral blood mononuclear cells will be isolated from the drawn peripheral blood. Using intra- and extracellular flowcytometry Vy9Vd2-T cells will be characterized phenotypically (APC markers: CD1d, CD40, CD80, CD83, CD86, HLA-DR; activation/memory markers: CD25, CD27, CD45RA, CD45RO, CCR7).
Occurrence of a febrile response | 2 days
  Patients will be requested to measure their temperature thrice daily during the 2 days following the first aminobisphosponate administration. This, because a relation between the occurrence of a febrile response upon aminobisphosponate administration and an activation and expansion of Vy9Vd2-T cells has been suggested.
Functional (IFN-γ, TNF-α, granzyme B) changes in the circulating pool of Vy9Vd2-T cells. | 5 weeks
  Peripheral blood mononuclear cells will be isolated from the drawn peripheral blood. Using intra- and extracellular flowcytometry Vy9Vd2-T cells will be characterized functionally (IFN-γ, TNF-α, granzyme B).

CONTACTS AND LOCATIONS:
Overall Officials: J J van der Vliet, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands